CLINICAL TRIAL: NCT07323615
Title: A Single-Center Randomized Controlled Trial Comparing the Efficacy and Safety of Naked-Eye Observation Versus Microscopic Magnification Observation in the Treatment of Skin Wounds
Brief Title: A Comparative Study of the Efficacy and Safety of Two Methods in the Treatment of Skin Wounds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Song Gu, Deputy Director for Administration, Trauma Center, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shanghai1st-SGu-1
Record Dates: First submitted 2025-12-10; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Wound Debridement
Keywords: skin wound; infection; debridement; microscope; therapeutic effect
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Debridement under microscopic magnification assistance plus Vacuum Sealing Drainage (VSD).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- naked-eye (No Intervention): Debridement under naked-eye observation plus Vacuum Sealing Drainage (VSD)
- microscopic (Experimental): Debridement under microscopic magnification assistance plus Vacuum Sealing Drainage (VSD).
  Interventions: Device: microscopic

INTERVENTIONS:
Device: microscopic — debridement with surgical microscope
  Arms: microscopic

SUMMARY:
This study will compare the experimental group (debridement assisted by surgical microscope + VSD) and the control group (debridement under naked-eye observation + VSD) in terms of the rate of change in BWAT scores at one week postoperatively when the VSD is removed, daily wound negative-pressure drainage volume and pain scores within the first postoperative week, and results of two wound bacterial cultures. The study aims to scientifically evaluate the difference in efficacy between microscope-assisted debridement and naked-eye debridement, with the goal of providing a reference for the clinical debridement treatment of skin wounds.

DETAILED DESCRIPTION:
Skin, which covers the body surface, is the outermost and largest organ of the human body. It is highly susceptible to various types of injuries, leading to acute or chronic wounds. Acute wounds typically result from sudden trauma, such as abrasions, friction injuries, cuts, or punctures, and are relatively easier to treat. Chronic wounds, on the other hand, refer to wounds that fail to achieve anatomical and functional integrity within the expected timeframe despite standardized and systematic treatment. Their pathogenesis is complex and often closely associated with multiple pathological factors such as infection, diabetic peripheral neuropathy and ischemic changes, persistent inflammatory responses, venous insufficiency, pressure injuries, and radiation damage. Such wounds are not only prolonged and recurrent, significantly impairing patients' quality of life, but also pose a major clinical challenge due to their difficulty in treatment and slow healing.

For skin wounds, the treatment principle is to perform thorough debridement first, followed by reconstructive surgery to cover the wound once infection is effectively controlled. Debridement is the core step in wound management, and its thoroughness directly impacts infection control, granulation tissue growth, and the final healing outcome. The 2023 Guidelines for the Diagnosis and Treatment of Chronic Refractory Wounds in Traumatic Orthopedics: Treatment Summary states that debridement, as the critical initial step in wound treatment, aims to remove necrotic tissue, reduce bioburden, control infection, and create favorable conditions for healing. The guidelines particularly emphasize adherence to the principle of "moderate debridement" , which involves thoroughly removing nonviable and heavily contaminated tissue while preserving as much viable tissue as possible to balance the completeness of wound bed preparation with the need for tissue preservation. Traditional debridement primarily relies on the surgeon's naked-eye observation and experience, which may fail to fully identify and remove all necrotic/infected tissue, micro-foreign bodies, and biofilms, or may lead to excessive debridement causing damage to healthy tissue. Both scenarios can impair wound bed preparation and ultimately affect the outcome of reconstructive surgery.

The surgical microscope is a commonly used device in trauma orthopedics and microsurgery, providing the surgeon with magnified, three-dimensional, and well-illuminated visual fields, mainly for the suturing and repair of delicate structures such as blood vessels and nerves. To date, there have been few reports on the use of surgical microscopes for skin wound debridement. Theoretically, with the aid of a microscope, clinicians could further enhance the discrimination between viable and necrotic tissue, achieving more precise and thorough debridement.

VSD (Vacuum Sealing Drainage) technology is an efficient drainage method that utilizes VSD materials and a semi-permeable membrane to isolate the wound from the external environment and promotes healing through continuous negative-pressure suction. The technique was first introduced by Dr. Fleischmann at Ulm University in Germany in 1992 and was introduced to China in 1994. The VSD negative-pressure closed drainage system consists of VSD material, a semi-permeable membrane, a three-way connector, and a negative-pressure suction device. It has been widely used in the treatment of skin wounds and can significantly improve local blood flow, reduce tissue edema, inhibit bacterial proliferation, and promote granulation tissue growth. Generally, one closed drainage session can maintain effective drainage for 5-7 days without requiring daily dressing changes.

The Bates-Jensen Wound Assessment Tool (BWAT) was developed by Bates-Jensen et al. in 1990 and revised in 2001. The revised BWAT includes two non-scored items (wound location and shape) and 13 scored items (size, depth, edges, undermining, necrotic tissue type and amount, exudate type and amount, periwound skin color, peripheral tissue edema and induration, granulation tissue, and epithelialization). The total score is the sum of the 13 item scores, with higher scores indicating more severe wound conditions. The validity and advantages of simplicity and speed of the BWAT have been confirmed in multiple clinical studies, providing objective and reliable data for assessing wound healing progress. Karahan tested the reliability and validity of the Turkish version of the BWAT, showing a content validity of 0.82 and a Cronbach's α coefficient of 0.85.

The surgical microscope offers advantages such as low cost, ease of operation, and integration into existing surgical workflows. A key foundation for the smooth implementation of this study is the full availability and routine use of internationally standardized, high-precision surgical microscope systems in the operating rooms of our hospital. This equipment is not temporarily acquired or specially introduced for this study but is an integral part of the standard operating room setup. Its performance parameters have been strictly calibrated and are maintained daily, fully meeting the technical requirements set by this study protocol. The devices are in good condition, regularly serviced and optically calibrated by professional engineers to ensure optimal imaging quality. Their stable yet flexible mounting systems accommodate different surgical positions and operator preferences. The surgical team is highly proficient in their operation, greatly facilitating the immediate initiation and efficient execution of the study protocol, thereby providing a solid guarantee for obtaining high-quality data within the planned timeframe.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged ≥18 years
2. Patients with chronic skin wounds requiring surgical debridement due to causes such as trauma, diabetes, venous ulcers, or pressure injuries
3. Patients whose systemic underlying medical conditions permit surgical tolerance
4. Patients who agree to participate in the clinical study and provide signed informed consent

Exclusion Criteria:

1. Presence of severe systemic immune diseases
2. Known allergy to any component of the Vacuum Sealing Drainage (VSD) dressing
3. Wounds with uncontrollable active major hemorrhage
4. Visible bone fragments or internal fixation materials within the wound
5. Pregnancy or lactation
6. Inability to cooperate with or complete follow-up

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
To compare the rate of change in wound scores between two methods of skin wound debridement. | one week
  the rate of change in wound scores= (BWAT score at 1-week post-debridement (VSD removal) - Pre-debridement BWAT score) / Pre-debridement BWAT score. The Bates-Jensen Wound Assessment Tool (BWAT) is a comprehensive, standardized instrument designed for the detailed assessment and documentation of wound characteristics. It is widely used by healthcare professionals, particularly in wound care, dermatology, and long-term care settings, to evaluate a variety of chronic wounds, including pressure injuries, venous stasis ulcers, diabetic foot ulcers, and surgical wounds. The strength of the BWAT lies in its structured approach. It assesses 13 key wound characteristics, each characteristic is scored from 1-5. The HIGHER the total score(13-65), the more severe the wound status.

SECONDARY OUTCOMES:
To compare the daily volume of wound negative pressure drainage between the two groups within one week postoperatively | one week
  Measure the volume of wound negative pressure drainage between the two groups everyday within one week postoperatively
To compare the daily pain scores of patients between the two groups within one week postoperatively | one week
  The Visual Analogue Scale (VAS) was used to record pain scores.
To compare the rate of conversion from positive to negative in wound bacterial culture between the two groups at one week postoperatively | two weeks
  Wound secretion bacterial cultures were performed both before and after the debridement procedure, each of which required approximately one week to obtain the results (positive or negative).
To compare the length of hospital stay between the two groups | through study completion, an average of 1 month
  The total number of days from hospital admission to discharge was calculated.

IPD SHARING:
Plan to Share IPD: Yes
individual participant data, as well as the study protocol, statistical analysis plan, and clinical study report.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Sharing will begin within 6 months after the publication of the main study results in a peer-reviewed journal, last for 5 years.
Access Criteria: Data will be made available to qualified researchers whose study proposals have been approved by an independent Data Access Committee for the purpose of independent verification or secondary meta-analysis.